CLINICAL TRIAL: NCT02775565
Title: Initial Experience With the AngioVac Venous Drainage Cannula and Cardiopulmonary Bypass Circuit: A Retrospective, Multi-Center Chart Review
Brief Title: Initial Experience With the AngioVac Venous Drainage Cannula
Status: Completed | Type: Observational
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PV-AV400
Record Dates: First submitted 2016-04-25; First posted 2016-05-17 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AngioVac

SUMMARY:
This is a retrospective, record-based study of approximately 100 patients across up to 12 centers within the United States. All patients who have been treated with the AngioVac Venous Drainage Cannula and the Extracorporeal Circuit will be considered for study participation. Eligible subject must meet all of the inclusion criteria and none of the exclusion criteria to be considered enrolled in the study. The purpose of the study is to describe initial experience with the AngioVac Venous Drainage Cannula and the Extracorporeal Circuit.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients treated at each study site between February 1, 2013 and February 28, 2015 will be included.

Exclusion Criteria:

* Patients treated with the AngioVac venous drainage system outside of those dates.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients treated at each study site between February 1, 2013 and February 28, 2015 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Detailing early clinical experience with the AngioVac Venous Drainage Cannula | Experience and success is determined immediately after the procedure is completed. No subject follow up data is collected and retrospective data will be reviewed.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Providence St. Joseph, Burbank, California
  - UCLA, Los Angeles, California
  - Sanford Research, Fargo, North Dakota
  - MUSC, Charleston, South Carolina
  - Swedish Health Services, Seattle, Washington